CLINICAL TRIAL: NCT04557878
Title: Role of Liquid Phase Concentrated Growth Factors vs. Hypertonic Dextrose Prolotherapy for Management of Patients With Disc Displacement Without Reduction (A Randomized Clinical Trial)
Brief Title: Role of Liquid Phase Concentrated Growth Factors vs. Hypertonic Dextrose Prolotherapy for Management of Patients With Disc Displacement Without Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPGF vs hypertonic dextrose
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Dextrose Solution (Experimental)
  Interventions: Drug: Hypertonic Dextrose Solution
- Liquid Phase Concentrated Growth Factor (LPCGFs) (Active Comparator)
  Interventions: Biological: Liquid Phase Concentrated Growth Factor (LPCGFs)

INTERVENTIONS:
Drug: Hypertonic Dextrose Solution — Patients in this group will receive an intra-articular injection of 12.5% hypertonic dextrose solution, once every month for three consecutive months, in conjugation with a maxillary CAD/CAM full-arch hard clear acrylic stabilization appliance.The point of needle entry will be 1 cm below the apex of the zygomatic arch and guided by ultrasound to ensure intra-articular injection in the superior joint space.
  Arms: Hypertonic Dextrose Solution
Biological: Liquid Phase Concentrated Growth Factor (LPCGFs) — Patients in this group will receive single intra-articular injection of LPCGF in conjugation with a maxillary CAD/CAM full-arch hard clear acrylic stabilization appliance.
  Arms: Liquid Phase Concentrated Growth Factor (LPCGFs)

SUMMARY:
Purpose of the study is to compare clinically, radiographically and biochemically the effect of intra- articular injection of hypertonic dextrose with a stabilization appliance and the intra- articular injection of 2 ml of liquid phase concentrated growth factor with a stabilization appliance as a prolotherapy for temporomandibular joint anterior disc displacement without reduction.

DETAILED DESCRIPTION:
Twenty four patients with anterior disc displacement without reduction will be selected from those attending the Prosthodontic Department, Faculty of Dentistry, Alexandria University and diagnosed clinically and by magnetic resonance imaging. Patients will be randomly assigned into 2 study groups each comprising 12 patients. Group I will receive an intra-articular injection of hypertonic dextrose in conjugation with a maxillary CAD/CAM full-arch hard clear acrylic stabilization appliance while group II will receive an intra-articular injection of LPCGF in conjugation with a maxillary CAD/CAM full-arch hard clear acrylic stabilization appliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful TMJ.
* Patients with limited mouth opening (MMO <40mm).
* Patients with anterior disc displacement without reduction confirmed by MRI.
* Presence of full or nearly full complement of natural teeth.
* Patients with angle class I occlusion.
* Patients with RCP not greater than 2mm and with no open bite.

Exclusion Criteria:

* Patients who have anterior disc dislocation with reduction detected by MRI.
* Inability or unwillingness to undergo magnetic resonance imaging (MRI) such as implanted electronic devices.
* Patients having uncontrolled systemic disease, hematologic or neurologic disorders or inflammatory diseases.
* Patients under anticoagulant drug therapy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum mouth opening | up to 6 months
  This will be evaluated using Helkimo Anamnestic index (Ai) which comprises the following classes: Ai0 - absence of subjective symptoms of dysfunction; AiI -mild symptoms, such as TMJ sounds, including clicking and crepitation, and feelings of stiffness or fatigue of the jaws; and AiII - severe symptoms of dysfunction, such as difficulty in opening the mouth wide, locking, luxations, pain on movement, and facial and jaw pain.
Disc-condyle relationship | 6 months
  This will be evaluated using magnetic resonance imaging (MRI) to assess the position of the articular disc and the condyle and the mandibular fossa
Myeloperoxidase enzyme activity | 6 months
  This will be evaluated by using Myeloperoxidase enzyme assay kits for detection and quantitation of myeloperoxidase activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam M. Bahgat, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Nadia R El-Helw, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Ahmed Abdelhamid, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Mohamed Fata, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Medhat Ashour, PhD, Study Director — High Institute of Public Health, Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt